CLINICAL TRIAL: NCT07015489
Title: A Prospective, Single-center Phase II Clinical Study of Concurrent Radiotherapy Following Induction Chemoimmunotherapy for Locally Advanced Esophageal Cancer
Brief Title: Concurrent Radiotherapy Following Induction Chemoimmunotherapy for Locally Advanced Esophageal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GXL-006
Record Dates: First submitted 2025-05-23; First posted 2025-06-11 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: ESCC
Keywords: induction immunochemotherapy
MeSH Terms: interventions — Induction Chemotherapy; Immunotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Induction therapy group (Experimental)
  Interventions: Drug: induction chemotherapy and immunotherapy

INTERVENTIONS:
Drug: induction chemotherapy and immunotherapy — All patients will first receive 2 cycles of induction chemoimmunotherapy, followed by radiotherapy. During radiotherapy, 2 concurrent cycles of chemoimmunotherapy will be administered. Afterward, maintenance immunotherapy will continue for up to one year.
  Chemotherapy regimen: Paclitaxel: 135 mg/m², Day 1, every 3 weeks (Q3W); Carboplatin: area under the curve (AUC) = 5, intravenous infusion over more than 30 minutes, Day 2, Q3W; Alternatively, Nedaplatin: 75 mg/m², Day 2, Q3W.
  Immunotherapy regimen: programmed death-1 (PD-1) inhibitor (e.g., Camrelizumab): Day 0, intravenous infusion, Q3W; Continued until disease progression (PD) or unacceptable toxicity, for a maximum duration of one year.
  Radiotherapy: Prescribed dose: 95% of the planning target volume (PTV) and planning target volume for nodal disease (PTV-nd) should receive 50-50.4 Gy over 25-28 fractions; Fraction dose range: 1.8-2.0 Gy per fraction, 5 days per week; External beam radiotherapy to the chest.

SUMMARY:
Esophageal cancer is one of the most common malignancies, and concurrent chemoradiotherapy (CRT) is the standard treatment for unresectable, locally advanced esophageal squamous cell carcinoma. In recent years, studies have suggested that combining immunotherapy with definitive CRT may further improve treatment outcomes. Currently, several clinical trials are underway to evaluate the efficacy of immunotherapy combined with chemotherapy (chemo) and radiotherapy in patients with unresectable, locally advanced esophageal cancer. The investigators plan to conduct a single-arm, prospective, single-center phase II clinical study to investigate the efficacy and safety of induction chemo and immunotherapy followed by concurrent radiotherapy (RT) in the treatment of locally advanced esophageal cancer. A total of 44 patients will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

1. The patient voluntarily agrees to participate in this study, has signed the informed consent form, demonstrates good compliance, and agrees to cooperate with follow-up.
2. Age ≥ 18 years, regardless of gender.
3. Histologically confirmed locally advanced esophageal squamous cell carcinoma, clinical stage II-IV and deemed unresectable (including unresectable cases, patients with surgical contraindications, or those who refuse surgery) based on the 8th edition of the American Joint Committee on Cancer (AJCC) staging system. Pre-treatment clinical staging: cT1N2-3M0, cT2-4bN0-3M0, or M1 limited to non-regional lymph node metastasis (excluding distant organ metastasis).
4. At least one measurable lesion as defined by Response Evaluation Criteria In Solid Tumors (RECIST) version 1.1.
5. No prior systemic antitumor therapy (including but not limited to systemic chemotherapy, radiotherapy, targeted therapy, immunotherapy, biologic therapy,local treatments, or other investigational treatments).
6. Eastern Cooperative Oncology Group (ECOG) performance status: 0-1.
7. Expected survival of ≥ 6 months.
8. Adequate function of major organs as defined below (use of any blood components or growth factors is not allowed within 2 weeks prior to screening):

absolute neutrophil count (ANC) ≥ 1.5 × 10⁹/L; Platelets ≥ 100 × 10⁹/L; Hemoglobin ≥ 100 g/L (female), ≥ 110 g/L (male); Serum albumin ≥ 2.8 g/dL; Total bilirubin ≤ 1.5 × upper limit of normal (ULN); alanine aminotransferase (ALT), aspartate aminotransferase (AST), and/or alkaline phosphatase (ALP) ≤ 2.5 × ULN; Serum creatinine ≤ 1.5 × ULN or creatinine clearance rate ≥ 60 mL/min (calculated using the Cockcroft-Gault formula); international normalized ratio (INR) and activated partial thromboplastin time (APTT) ≤ 1.5 × ULN (patients receiving stable doses of anticoagulants such as low molecular weight heparin or warfarin with INR within the expected therapeutic range of the anticoagulant may be eligible for screening).

Female participants: All women of childbearing potential must have a negative serum pregnancy test during screening and must agree to use reliable contraception from the time of signing the informed consent form until 3 months after the last dose.

Exclusion Criteria:

1. History of esophageal cancer surgery.
2. History of fistula caused by primary tumor invasion.
3. High risk of gastrointestinal bleeding, esophageal fistula, or esophageal perforation.
4. Poor nutritional status, with ≥10% body weight loss within 2 months prior to screening and no significant improvement after nutritional intervention.
5. Major surgery or severe trauma within 4 weeks prior to first administration of the investigational drug.
6. Presence of uncontrollable pleural effusion, pericardial effusion, or ascites requiring repeated drainage.
7. Prior or ongoing treatment with any of the following:

   1. Anti-programmed death-1 (PD-1) or anti-programmed death-ligand 1 (PD-L1) antibody therapy, chemotherapy, radiotherapy, or targeted therapy.
   2. Use of any investigational drug within 4 weeks prior to first administration of the study drug.
   3. Systemic use of corticosteroids (daily dose >10 mg prednisone or equivalent) or other immunosuppressive agents within 2 weeks prior to first dose of the study drug, except for local esophageal inflammation, prophylaxis against allergies, or antiemetic use. Special circumstances require consultation with the sponsor. Inhaled or topical steroids and adrenal hormone replacement at >10 mg/day prednisone-equivalent are allowed in the absence of active autoimmune disease.
8. Receipt of anti-tumor vaccines or live vaccines within 4 weeks prior to first dose of the study drug.
9. Presence or history of any active autoimmune disease (e.g., interstitial pneumonitis, uveitis, colitis, hepatitis, hypophysitis, vasculitis, myocarditis, nephritis, hyperthyroidism, or hypothyroidism); exceptions include vitiligo, childhood asthma/allergies now resolved without intervention, autoimmune hypothyroidism on stable thyroid hormone replacement, and type I diabetes mellitus on stable insulin regimen.
10. History of immunodeficiency, including human immunodeficiency virus (HIV) positive status or other acquired or congenital immunodeficiency diseases, or history of organ or allogeneic bone marrow transplantation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | From treatment initiation through study completion (up to 3 years)
  The time from the start of treatment to tumor progression (of any form) or death from any cause.

SECONDARY OUTCOMES:
OS (overall survival) | From treatment initiation through study completion (up to 3 years)
Adverse Event (AE) | Up to 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No